CLINICAL TRIAL: NCT00183248
Title: Pilot Study Using Donor Stem Cells and Campath-1H to Induce Renal Transplant Tolerance (ITN022ST)
Brief Title: Using Donor Stem Cells and Alemtuzumab to Prevent Organ Rejection in Kidney Transplant Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Principal Investigator, George W. Burke, Professor of Surgery, National Institute of Allergy and Infectious Diseases (NIAID)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DAIT ITN022ST
Record Dates: First submitted 2005-09-11; First posted 2005-09-16 (Estimated); Results first posted 2012-06-21 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Kidney Transplantation; Kidney Disease; Kidney Failure
Keywords: kidney; kidney transplant; kidney transplantation; transplant; transplantation; renal; renal transplant; renal transplantation; kidney disease; chronic; renal failure; kidney failure
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency; Bronchiolitis Obliterans Syndrome | interventions — Alemtuzumab; Mycophenolic Acid; Sirolimus; Tacrolimus; Kidney Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DBMCs (Experimental): Kidney transplantation, followed by immunotherapy given along with kidney donor Donor bone Bone marrow Marrow stem cell Cells (DBMCs) infusions
  Interventions: Drug: Alemtuzumab; Drug: Mycophenolate mofetil; Drug: Sirolimus; Drug: Tacrolimus; Procedure: Donor bone marrow stem cell infusion; Procedure: Kidney transplant
- Control Group (Active Comparator): Kidney transplantation, followed by immunotherapy
  Interventions: Drug: Alemtuzumab; Drug: Mycophenolate mofetil; Drug: Sirolimus; Drug: Tacrolimus; Procedure: Kidney transplant

INTERVENTIONS:
Drug: Alemtuzumab — Immunosuppressant; 2 doses of drug by intravenous (IV) infusion on Days 0 and 4
  Other Names: Campath
Drug: Mycophenolate mofetil — Immunosuppressant; oral daily dose starting Day 0 until withdrawal or end of the study
  Other Names: Cellcept
Drug: Sirolimus — Immunosuppressant; oral daily dose starting between Months 4 and 6 post-transplant until withdrawal or end of the study
  Other Names: rapamycin, Rapamune
Drug: Tacrolimus — Immunosuppressant; daily dose starting Day 1 until withdrawal or end of the study
  Other Names: FK-506
Procedure: Donor bone marrow stem cell infusion — 2 doses of kidney donor's bone marrow stem cells by IV infusion on Day 5 and sometime between Months 4 and 6
  Arms: DBMCs
Procedure: Kidney transplant — Occurs at study entry

SUMMARY:
Alemtuzumab is a man-made antibody used to treat certain blood disorders. This study will evaluate treatment of kidney transplant recipients with alemtuzumab and other immune system suppressing medications with or without infusions of bone marrow stem cells from the kidney donor. The purpose of this study is to find out which strategy is more effective in preventing organ rejection and maintaining patient health.

DETAILED DESCRIPTION:
Organ transplantation is a common procedure in hospitals, but organ rejection and serious side effects are potential problems for the patient. Mycophenolate mofetil, sirolimus, and tacrolimus are drugs used to decrease immune system activity in people who have received organ transplants so that the new organ will not be rejected. Alemtuzumab is a monoclonal antibody that binds to and depletes excess T cells in the bone marrow of leukemia patients. In this study, alemtuzumab will be used to destroy the recipient's white blood cells (WBCs) at the time of transplantation. It is hoped that WBCs produced after alemtuzumab administration will recognize the transplanted liver as "self" and will not attack the new kidney.

To further assist the immune system in accepting the donor kidney, some patients in this study will also receive two infusions of bone marrow stem cells from the kidney donor. Bone marrow stem cells are adult blood cells from which other specialized blood cells, such as T cells, develop. Treatment with these cells is believed to create a state of "chimerism" in the body, where the immune cells of both the donor and recipient can coexist and tolerate the presence of a donor organ. This study will evaluate the safety and effectiveness of an antirejection regimen including alemtuzumab and other immunosuppressive medications and donor bone marrow stem cell infusions in patients undergoing kidney transplantation.

This study will last 3 years. Participants will be randomly assigned to receive either the full immunosuppressive therapy and donor bone marrow stem cell infusions (Group 1) or immunosuppressive therapy alone (Group 2). Patients will undergo kidney transplantation at the start of the study on Day 0. Patients will receive inpatient infusions of alemtuzumab on Days 0 and 4. Starting on Day 0, patients will begin taking mycophenolate mofetil; starting on Day 1, patients will also begin taking tacrolimus. On Day 5, patients in Group 1 will receive their first of 2 infusions of purified stem cells taken from the kidney donor's bone marrow; their second infusion of stem cells will occur sometime between Months 4 and 6 post-transplant.

Beginning between Months 4 and 6 post-transplant, all participants will begin receiving low-dose maintenance immunosuppressive therapy with sirolimus, as is typical for post-transplant antirejection therapy. One year post-transplant, patients will be evaluated for the potential to withdraw some or all of this maintenance immunotherapy. Participants will be monitored for 3 years post-transplant. Urine collection will occur at Week 1 and Months 1, 3, 6, and 9. At Months 12, 24, and 30, participants will undergo kidney biopsies. Blood collection will occur at regular intervals for laboratory tests to evaluate the immune system's response to the transplanted kidney.

ELIGIBILITY:
Inclusion Criteria:

* Weight greater than 40 kg (88.2 lbs)
* Will be receiving a living-related (1-haplotype-matched donor/recipient) primary kidney allograft
* Negative B-cell and T-cell cytotoxic and flow cytometry crossmatch (1-haplotype-matched donor/recipient pairs with a minimum of 1 HLA DR 1A and 1B locus in common and panel-reactive antibodies [PRA] of less than 10%)
* Normal echocardiogram (ECG) with an ejection fraction of greater than 50%
* Received full course of vaccination for hepatitis B virus (HBV), completed at least 6 weeks before transplantation, OR has naturally acquired immunity
* Willing to comply with the study visits
* Willing to use acceptable forms of contraception

Exclusion Criteria:

* Previously received or is receiving an organ transplant other than a kidney
* Receiving an ABO (blood type) incompatible donor kidney
* Human Immunodeficiency Virus (HIV) infected
* Antibody positive for hepatitis C virus (HCV)
* Surface antigen positive for hepatitis B virus (HBV)
* Recipient or donor is positive for tuberculosis (TB), under treatment for suspected TB, or previously exposed to TB (positive Mantoux test)
* Current cancer or a history of cancer within the 5 years prior to study entry. Patients who have had successfully treated nonmetastatic basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix are not excluded.
* Significant liver disease, defined as having continuously elevated aspartate aminotransferase (AST SGOT) or alanine aminotransferase (ALT SGPT) levels greater than 3 times the upper value of the normal range within 28 days prior to study entry
* Uncontrolled concomitant infections, severe diarrhea, vomiting, active upper gastrointestinal tract malabsorption, active peptic ulcer, or any other unstable medical condition that could interfere with this study
* Currently receiving an investigational drug or received an investigational drug within 30 days prior to transplant
* Currently receiving any immunosuppressive agent
* Anticipated contraindication to taking medications orally or via nasogastric tube by the morning of Day 2 following completion of the transplant procedure
* Require certain medications
* Known hypersensitivity to any of the study medications, thymoglobulin daclizumab, or corticosteroids
* Certain screening laboratory values. More information on this criterion can be found in the protocol.
* Any form of substance abuse, psychiatric disorder, or other condition that, in opinion of the investigator, may interfere with the study
* Anticipated contraindication to tacrolimus administration for longer than 5 days post-transplant
* Currently undergoing peritoneal dialysis
* PRA value less than 10% at any time prior to study entry
* Graves disease. Patients with Graves disease adequately treated with radioiodine ablative therapy are not excluded.
* Cytomegalovirus (CMV) or Epstein-Barr virus (EBV) negative kidney recipient receiving a kidney from a CMV or EBV positive donor
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George W. Burke, III, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

REFERENCES:
- [Derived] Ciancio G, Sageshima J, Akpinar E, Gaynor JJ, Chen L, Zarak A, Hanson L, Tueros L, Guerra G, Mattiazzi A, Kupin W, Roth D, Ricordi C, Burke GW 3rd. A randomized pilot study of donor stem cell infusion in living-related kidney transplant recipients receiving alemtuzumab. Transplantation. 2013 Nov 15;96(9):800-6. doi: 10.1097/TP.0b013e3182a0f68c. PMID 23903014
- See also: Click here for the Immune Tolerance Network Web site — http://www.immunetolerance.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One center in the United States enrolled nine subjects who were recipients of living-related (1-haplotype-matched) donor kidney transplants between September 2004 and November 2006.
Pre-assignment Details: Participants underwent procedures at screening to establish inclusion/exclusion criteria.
Groups:
- DBMCs: Recipients of 1-haplotype human leukocyte antigen (HLA) matched living-donor related kidney transplantation were randomized to receive (CD34+ stem cell purified) Donor-specific Bone Marrow Cells (DBMCs). Induction therapy included alemtuzumab and steroid-free dose maintenance immunosuppression consisting of mycophenolate mofetil, tacrolimus and sirolimus. Refer to section titled 'Detailed Description' for additional treatment information.
- Control Group: Recipients of 1-haplotype human leukocyte antigen (HLA) matched living-donor related kidney transplantation were randomized to receive induction therapy with alemtuzumab and steroid-free dose maintenance immunosuppression consisting of mycophenolate mofetil, tacrolimus and sirolimus. Refer to section titled 'Detailed Description' for additional treatment information.
Period: Overall Study
Arm/Group | DBMCs | Control Group
Started | 4 | 5
Completed | 3 | 4
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Focal glomerulosclerosis proteinuria | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DBMCs | Control Group | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 41.0 (12.0) | 41.8 (7.9) | 41.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Participant Survival at One Year Post Kidney Transplant
Time Frame: One year post kidney transplant
Population: Intent-to-Treat
Measure: Number; unit: participants
Arm/Group | DBMCs | Control Group
Number analyzed (Participants) | 4 | 5
participants | 4 | 5

2. Primary Outcome: Overall Kidney Graft Survival at One Year Post-Transplant
Description: Number of participants that did not experience kidney graft failure[1] at one year post-transplant
  [1]Graft failure is defined as the institution of chronic dialysis (at least 6 consecutive weeks, excluding participants with delayed graft function), transplant nephrectomy, or retransplantation.
Time Frame: One year post kidney transplant
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | DBMCs | Control Group
Number analyzed (Participants) | 4 | 5
participants | 4 | 5

3. Secondary Outcome: Participant Survival at Three Years Post Kidney Transplant
Time Frame: Three years post kidney transplant
Population: Intent-to-Treat
Measure: Number; unit: participants
Arm/Group | DBMCs | Control Group
Number analyzed (Participants) | 4 | 5
participants | 4 | 5

4. Secondary Outcome: Graft Survival at Three Years Post-Transplant
Description: Number of participants that did not experience kidney graft failure[1] at three years post-transplant
  [1]Graft failure is defined as the institution of chronic dialysis (at least 6 consecutive weeks, excluding participants with delayed graft function), transplant nephrectomy, or retransplantation.
Time Frame: Three years post kidney transplant
Population: Intent-to-Treat
Measure: Number; unit: participants
Arm/Group | DBMCs | Control Group
Number analyzed (Participants) | 4 | 5
participants | 4 | 5

5. Secondary Outcome: Number of Kidney Biopsy-proven Acute Rejection
Description: Biopsy-proven acute renal (kidney) rejection[1,2].
  1. Diagnosis of acute rejection was made by renal biopsy using the Banff 97 criteria. The Banff 97 diagnostic category for renal allograft biopsies is an international standardized histopathological classification. Acute rejection is defined by a renal biopsy demonstrating a Banff 97 classification of Grade IA or greater, with higher scores indicating more severe rejection[2]
  2. Ref: Racusen LC et al. The Banff 97 working classification of renal allograft pathology. Kidney Int, 55: 713-723, 1999
Time Frame: Three years post kidney transplant
Population: Participants who experienced an acute rejection
Measure: Number; unit: Rejection Events
Arm/Group | DBMCs | Control Group
Number analyzed (Participants) | 1 | 1
Rejection Events | 1 | 1

6. Secondary Outcome: Number of Chronic Allograft Nephropathies
Description: Number of chronic allograft nephropathies[1,2,3] at 3 years post kidney transplant.
  1. Chronic allograft nephropathy is defined as renal biopsies with Banff 97 Grade I or greater[2] with higher numeric scores indicating more severe nephropathy
  2. The Banff 97 diagnostic category for renal allograft biopsies is an international standardized histopathological classification[3]
  3. Reference: Racusen LC, Solez K, Colvin RB et al. The Banff 97 working classification of renal allograft pathology. Kidney Int, 55: 713-723, 1999
Time Frame: Three years post kidney transplant
Population: Participants who experienced nephropathies
Measure: Number; unit: Nephropathy Events
Arm/Group | DBMCs | Control Group
Number analyzed (Participants) | 4 | 1
Nephropathy Events | 6 | 2

7. Secondary Outcome: Number of Graft-versus-host Disease (GVHD) Events
Description: A disease caused when cells from a donated stem cell graft attack the normal tissue of the transplant patient. Symptoms include jaundice, skin rash or blisters, a dry mouth, or dry eyes. Also called graft-versus-host disease.
Time Frame: Three years post kidney transplant
Population: Intent-to-Treat
Measure: Number; unit: GVHD Events
Arm/Group | DBMCs | Control Group
Number analyzed (Participants) | 4 | 5
GVHD Events | 0 | 0

ADVERSE EVENTS:
Arm/Group | DBMCs | Control Group
Serious Adverse Events (participants affected / at risk) | 4/4 | 3/5
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DBMCs (N=4) | Control Group (N=5)
Chest pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Kidney transplant rejection (Immune system disorders) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Drug toxicity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 3 (12) | 2 (2)
Glomerulonephritis membranoproliferative (Renal and urinary disorders) | 1 (1) | 0 (0)
Mesangioproliferative glomerulonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DBMCs (N=4) | Control Group (N=5)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Palatal oedema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Face oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 3 (4) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Body tinea (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (5) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (3)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 3 (3)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 0 (0)
Red blood cell count decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 3 (4) | 2 (3)
Menorrhagia (Reproductive system and breast disorders) | 1 (3) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tonsillar ulcer (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2)
Hypertension (Vascular disorders) | 2 (3) | 4 (6)

LIMITATIONS AND CAVEATS:
In July 2007 after the trial had been enrolling for approximately 42 months, enrollment was stopped at the current number of nine subjects due to time and resource constraints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No